CLINICAL TRIAL: NCT03282240
Title: Safety and Immunogenicity of High-Dose Quadrivalent Influenza Vaccine Administered by Intramuscular Route in Participants Aged 65 Years and Older
Brief Title: Safety and Immunogenicity of High-Dose Quadrivalent Influenza Vaccine in Participants ≥65 Years in the US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QHD00013; U1111-1183-5556 (Other: World Health Organization Universal Trial Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: QHD00013 was a phase III, randomized, modified double-blind, active-controlled, multi-center trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: QHD00013 was a modified double-blind trial with an unblinded administrator used at each trial site. The administrator was not involved in any of the blinded study assessments (e.g., safety).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- QIV-HD (Experimental): Participants randomized to receive a single injection of 0.7 mL QIV-HD by intramuscular (IM) route at Day 0.
  Interventions: Biological: QIV-HD
- TIV-HD1 (Licensed TIV-HD1) (Active Comparator): Participants randomized to receive a single injection of 0.5 mL licensed TIV-HD1 by IM route at Day 0.
  Interventions: Biological: Licensed TIV-HD1
- TIV-HD2 (Investigational TIV-HD2) (Active Comparator): Participants randomized to receive a single injection of 0.5 mL investigational TIV-HD2 by IM route at Day 0.
  Interventions: Biological: Investigational TIV-HD2

INTERVENTIONS:
Biological: QIV-HD — 0.7 mL-dose was administered intramuscularly (IM) into the upper arm area.
  Other Names: High-dose quadrivalent influenza vaccine
  Arms: QIV-HD
Biological: Licensed TIV-HD1 — 0.5 mL-dose was administered IM into the upper arm area.
  Other Names: High-dose trivalent influenza vaccine
  Arms: TIV-HD1 (Licensed TIV-HD1)
Biological: Investigational TIV-HD2 — 0.5 mL-dose was administered IM into the upper arm area.
  Other Names: High-dose trivalent influenza vaccine (alternate B strain)
  Arms: TIV-HD2 (Investigational TIV-HD2)

SUMMARY:
This randomized, modified double-blind, active-controlled, multi-center trial assessed the safety and immunogenicity of the high-dose quadrivalent influenza vaccine (QIV-HD) compared to either the licensed or investigational high-dose trivalent influenza vaccine (TIV-HD) in adults.

DETAILED DESCRIPTION:
This randomized, modified double-blind, active-controlled, multi-center trial was conducted in healthy adults (greater than and equal to [>=] 65 years) to assess the safety and immunogenicity (geometric mean titers and seroconversion for the 4 virus strains at 28 days post vaccination) of the QIV-HD compared to one of the TIV-HDs containing either the B strain from the primary lineage (TIV-HD1; licensed vaccine [Fluzone® High-Dose] for the 2017-2018 Northern Hemisphere [NH] influenza season) or the B strain from the alternate lineage (TIV-HD2, investigational TIV-HD containing an alternate B strain).

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 65 years on the day of inclusion.
* Informed consent form had been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation at the time of trial enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2.
* Previous vaccination against influenza (in the preceding 6 months) with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on investigator's judgment.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Alcohol or substance abuse that, in the opinion of the investigator, might interfere with the trial conduct or completion.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Identified as an Investigator or employee of the Investigator or trial center with direct involvement in the proposed trial, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed trial.
* Personal or family history of Guillain-Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy and participants who have a history of neoplastic disease and have been disease free for >= 5 years).
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0°C [>= 100.4°F]). A prospective participant should not be included in the trial until the condition has resolved or the febrile event had subsided.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2670 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (36):
- United States (36):
  - Sanofi Pasteur Investigational Site 037, Anaheim, California
  - Sanofi Pasteur Investigational Site 029, Redding, California
  - Sanofi Pasteur Investigational Site 003, San Diego, California
  - Sanofi Pasteur Investigational Site 016, Colorado Springs, Colorado
  - Sanofi Pasteur Investigational Site 035, Milford, Connecticut
  - Sanofi Pasteur Investigational Site 031, Hollywood, Florida
  - Sanofi Pasteur Investigational Site 009, Jacksonville, Florida
  - Sanofi Pasteur Investigational Site 017, Jacksonville, Florida
  - Sanofi Pasteur Investigational Site 030, Stockbridge, Georgia
  - Sanofi Pasteur Investigational Site 010, Boise, Idaho
  - Sanofi Pasteur Investigational Site 034, Meridian, Idaho
  - Sanofi Pasteur Investigational Site 021, Council Bluffs, Iowa
  - Sanofi Pasteur Investigational Site 023, Wichita, Kansas
  - Sanofi Pasteur Investigational Site 028, Wichita, Kansas
  - Sanofi Pasteur Investigational Site 012, Bardstown, Kentucky
  - Sanofi Pasteur Investigational Site 018, Metairie, Louisiana
  - Sanofi Pasteur Investigational Site 026, Biloxi, Mississippi
  - Sanofi Pasteur Investigational Site 014, St Louis, Missouri
  - Sanofi Pasteur Investigational Site 011, Omaha, Nebraska
  - Sanofi Pasteur Investigational Site 024, Las Vegas, Nevada
  - Sanofi Pasteur Investigational Site 008, Rochester, New York
  - Sanofi Pasteur Investigational Site 005, Wilmington, North Carolina
  - Sanofi Pasteur Investigational Site 036, Winston-Salem, North Carolina
  - Sanofi Pasteur Investigational Site 004, Cleveland, Ohio
  - Sanofi Pasteur Investigational Site 015, Oklahoma City, Oklahoma
  - Sanofi Pasteur Investigational Site 013, Warwick, Rhode Island
  - Sanofi Pasteur Investigational Site 033, Mt. Pleasant, South Carolina
  - Sanofi Pasteur Investigational Site 001, Nashville, Tennessee
  - Sanofi Pasteur Investigational Site 002, Dallas, Texas
  - Sanofi Pasteur Investigational Site 025, Tomball, Texas
  - Sanofi Pasteur Investigational Site 027, Salt Lake City, Utah
  - Sanofi Pasteur Investigational Site 006, Salt Lake City, Utah
  - Sanofi Pasteur Investigational Site 019, Salt Lake City, Utah
  - Sanofi Pasteur Investigational Site 020, South Jordan, Utah
  - Sanofi Pasteur Investigational Site 022, West Jordan, Utah
  - Sanofi Pasteur Investigational Site 038, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Chang LJ, Meng Y, Janosczyk H, Landolfi V, Talbot HK; QHD00013 Study Group. Safety and immunogenicity of high-dose quadrivalent influenza vaccine in adults >/=65 years of age: A phase 3 randomized clinical trial. Vaccine. 2019 Sep 16;37(39):5825-5834. doi: 10.1016/j.vaccine.2019.08.016. Epub 2019 Aug 17. PMID 31431411
- See also: Related info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were screened in 35 centers in the Unites States (US) from 08 September 2017 to 15 September 2017.
Pre-assignment Details: A total of 2670 participants were randomized in the study.
Groups:
- High-Dose Quadrivalent Influenza Vaccine (QIV-HD): Participants randomized to receive a single injection of 0.7 mL high dose quadrivalent influenza vaccine (QIV-HD) by intramuscular (IM) route at Day 0.
- High-Dose Trivalent Influenza Vaccine (Licensed TIV-HD1): Participants randomized to receive a single injection of 0.5 mL licensed high dose trivalent influenza vaccine (TIV-HD1) by IM route at Day 0.
- High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2): Participants randomized to receive a single injection of 0.5 mL investigational high dose trivalent influenza vaccine with alternate B strain (TIV-HD2) by IM route at Day 0.
Period: Overall Study
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccine (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Started | 1777 | 443 | 450
Completed | 1767 | 440 | 447
Not Completed | 10 | 3 | 3
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Protocol Deviation | 4 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants for whom a vaccine group was allocated.
Groups:
- High-Dose Quadrivalent Influenza Vaccine (QIV-HD): Participants randomized to receive a single injection of 0.7 mL QIV-HD by IM route at Day 0.
- High-Dose Trivalent Influenza Vaccine (Licensed TIV-HD1): Participants randomized to receive a single injection of 0.5 mL licensed TIV-HD1 by IM route at Day 0.
- High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2): Participants randomized to receive a single injection of 0.5 mL investigational TIV-HD2 by IM route at Day 0.
- Total: Total of all reporting groups
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccine (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2) | Total
Number analyzed (Participants) | 1777 | 443 | 450 | 2670
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (5.63) | 72.8 (5.79) | 73.2 (5.49) | 73.0 (5.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1027 | 268 | 252 | 1547
  Male | 750 | 175 | 198 | 1123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 2 | 3 | 14
  Asian | 13 | 2 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 1 | 6
  Black or African American | 123 | 41 | 35 | 199
  White | 1618 | 395 | 402 | 2415
  More than one race | 6 | 1 | 2 | 9
  Unknown or Not Reported | 4 | 1 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Antibodies Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: GMTs of anti-influenza antibodies were measured using an hemagglutination inhibition (HAI) assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). For each A strain, the comparison was made with the pooled TIV-HD groups. For each B strain, the comparison was made with the TIV-HD group containing the corresponding B strain. TIV-HD 1 did not contain B2 strain; TIV-HD2 did not contain B1 strain.
Time Frame: Day 28 post-vaccination
Population: Per-protocol analysis set (PPAS): all randomized participants who received at least 1 dose of trial vaccine & had a post-vaccination blood sample HAI result for at least 1 strain, with no relevant protocol deviations. Here, 'number analyzed' = participants with available data for each category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1): Participants randomized to receive a single injection of 0.5 mL licensed TIV-HD1 by IM route at Day 0.
- High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled): Participants randomized to receive either a single injection of 0.5 mL licensed TIV-HD1 or investigational TIV-HD2 by IM route at Day 0.
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2) | High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled)
Number analyzed (Participants) | 1680 | 423 | 430 | 853
titers (1/dilution)
  A/H1N1 | 312 [292 to 332] | 387 [339 to 442] | 362 [317 to 413] | 374 [341 to 411]
  A/H3N2: number analyzed (Participants) | 1679 | 423 | 430 | 853
  A/H3N2 | 563 [525 to 603] | 588 [513 to 673] | 600 [524 to 687] | 594 [540 to 653]
  B Victoria: number analyzed (Participants) | 1680 | 423 | 0 | 0
  B Victoria | 516 [488 to 545] | 476 [426 to 532] |  |
  B Yamagata: number analyzed (Participants) | 1680 | 0 | 430 | 0
  B Yamagata | 578 [547 to 612] |  | 580 [519 to 649] |
Statistical Analysis 1: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1); B Victoria: The 2-sided 95% confidence interval (CI) was based on the Student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results; Test type: Non-Inferiority — Non-inferiority of GMTs was concluded if the lower limit of the 2-sided 95% CI of the ratio of GMTs between groups is > 0.667 for each of the comparisons; GMT Ratio (QIV-HD/TIV-HDs) = 1.08, 95% CI 2-sided [0.958 to 1.224]
Statistical Analysis 2: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2); B Yamagata: The 2-sided 95% CI was based on the Student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT Ratio (QIV-HD/TIV-HDs) = 1.00, 95% CI 2-sided [0.881 to 1.129]
Statistical Analysis 3: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled); A/H1N1: The 2-sided 95% CI was based on the Student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT Ratio (QIV-HD/TIV-HDs) = 0.83, 95% CI 2-sided [0.744 to 0.932]
Statistical Analysis 4: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled); A/H3N2: The 2-sided 95% CI was based on the Student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMT Ratio (QIV-HD/TIV-HDs) = 0.95, 95% CI 2-sided [0.842 to 1.066]

2. Primary Outcome: Percentage of Participants Achieving Seroconversion Against Antigens Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). Seroconversion was defined as either a HAI titer less than (<) 10 (1/dilution) at Day 0 and post-injection titer greater than or equal to (>=) 40 (1/dilution) at Day 28, or HAI titer >=10 (1/dilution) at Day 0 and a >=4-fold increase in HAI titer (1/dilution) at Day 28. For each A strain, the comparison was made with the pooled TIV-HD groups. For each B strain, the comparison was made with the TIV-HD group containing the corresponding B strain. TIV-HD 1 did not contain B2 strain; TIV-HD2 did not contain B1 strain.
Time Frame: Day 28 post-vaccination
Population: Analysis was performed on PPAS. Here, 'number analyzed' = participants with available data for each category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2) | High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled)
Number analyzed (Participants) | 1680 | 423 | 430 | 853
percentage of participants
  A/H1N1: number analyzed (Participants) | 1669 | 420 | 428 | 848
  A/H1N1 | 50.4 [48.0 to 52.8] | 56.2 [51.3 to 61.0] | 51.2 [46.3 to 56.0] | 53.7 [50.2 to 57.1]
  A/H3N2: number analyzed (Participants) | 1668 | 420 | 428 | 848
  A/H3N2 | 49.8 [47.3 to 52.2] | 52.9 [48.0 to 57.7] | 48.1 [43.3 to 53.0] | 50.5 [47.1 to 53.9]
  B Victoria: number analyzed (Participants) | 1669 | 421 | 0 | 0
  B Victoria | 36.5 [34.2 to 38.9] | 39.0 [34.3 to 43.8] |  |
  B Yamagata: number analyzed (Participants) | 1669 | 0 | 428 | 0
  B Yamagata | 46.6 [44.2 to 49.0] |  | 48.4 [43.5 to 53.2] |
Statistical Analysis 1: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1); B Victoria: The 2-sided 95% CI for the difference is based on the Wilson score method without continuity correction; Test type: Non-Inferiority — Non-inferiority in seroconversion was concluded if the lower limit of the 2-sided 95% CI of the differences of seroconversion rates between groups is > -10%; Difference in Percentage = -2.41, 95% CI 2-sided [-7.66 to 2.70]
Statistical Analysis 2: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2); B Yamagata: The 2-sided 95% CI for the difference is based on the Wilson score method without continuity correction; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in Percentage = -1.75, 95% CI 2-sided [-7.04 to 3.53]
Statistical Analysis 3: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled); A/H3N2: The 2-sided 95% CI for the difference is based on the Wilson score method without continuity correction; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in Percentage = -0.71, 95% CI 2-sided [-4.83 to 3.42]
Statistical Analysis 4: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines Pooled (TIV-HDs Pooled); A/H1N1: The 2-sided 95% CI for the difference is based on the Wilson score method without continuity correction; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in Percentage = -3.27, 95% CI 2-sided [-7.37 to 0.86]

3. Secondary Outcome: GMTs of B Strains Influenza Antibodies Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: A/H1N1 (A1), A/H3N2 (A2), B Victoria lineage (B1), and B Yamagata lineage (B2). For each B strain, the immunogenicity of QIV-HD was compared to that of TIV-HD group which contains the corresponding B strain. TIV-HD1 did not contain B2 strain; TIV-HD2 did not contain B1 strain.
Time Frame: Day 28 post-vaccination
Population: Analysis was performed on full analysis set (FAS) that consisted who received at least 1 dose of a trial vaccine and had a post-vaccination blood sample HAI result for at least 1 strain. Participants were analyzed according to the vaccine group to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1763 | 439 | 446
titers (1/dilution)
  B Victoria: number analyzed (Participants) | 1763 | 0 | 446
  B Victoria | 515 [488 to 543] |  | 253 [227 to 283]
  B Yamagata: number analyzed (Participants) | 1763 | 439 | 0
  B Yamagata | 573 [542 to 605] | 280 [249 to 316] |
Statistical Analysis 1: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1); The 2-sided 95% CI is based on the Student t-distribution of logarithmic transformation of the individual titers. Antilog transformations were applied to the results; Test type: Superiority — Superiority in GMTs was observed if the lower limit of the 2-sided 95% CI of the ratio of GMTs between groups was > 1.5 for comparison group; GMT Ratio (QIV-HD/TIV-HDs) = 2.04, 95% CI 2-sided [1.804 to 2.315]
Statistical Analysis 2: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2); [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; GMT Ratio (QIV-HD/TIV-HDs) = 2.03, 95% CI 2-sided [1.802 to 2.288]

4. Secondary Outcome: GMT Ratios of Influenza Antibodies Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: GMTs of anti-influenza antibodies using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). Geometric Mean Titers Ratios (GMTRs) were calculated as the ratio of GMTs post vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Analysis was performed on PPAS. Here, 'number analyzed' = participants with available data for each category.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1680 | 423 | 430
ratio
  A/H1N1: Day28/Day 0: number analyzed (Participants) | 1669 | 420 | 428
  A/H1N1: Day28/Day 0 | 4.38 [4.11 to 4.66] | 5.57 [4.85 to 6.39] | 4.76 [4.16 to 5.44]
  A/H3N2: Day28/Day 0: number analyzed (Participants) | 1668 | 420 | 428
  A/H3N2: Day28/Day 0 | 4.65 [4.35 to 4.98] | 4.82 [4.24 to 5.48] | 4.94 [4.32 to 5.65]
  B Victoria: Day28/Day 0: number analyzed (Participants) | 1669 | 421 | 428
  B Victoria: Day28/Day 0 | 3.17 [2.99 to 3.35] | 3.35 [2.99 to 3.76] | 1.65 [1.52 to 1.78]
  B Yamagata: Day28/Day 0: number analyzed (Participants) | 1669 | 421 | 428
  B Yamagata: Day28/Day 0 | 3.82 [3.62 to 4.03] | 1.86 [1.73 to 2.02] | 3.82 [3.43 to 4.24]

5. Secondary Outcome: Percentage of Participants Achieving Seroconversion Against Antigens of B Strains After Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: Seroconversion was defined as either a HAI titer <10 (1/dilution) at Day 0 and post-injection titer >=40 (1/dilution) at Day 28, or HAI titer >=10 (1/dilution) at Day 0 and a >=4-fold increase in HAI titer (1/dilution) at Day 28.
Time Frame: Day 28 post-vaccination
Population: Analysis was performed on FAS. Here, 'number analyzed' = participants with available data for each category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1763 | 439 | 446
percentage of participants
  B Victoria: number analyzed (Participants) | 1751 | 0 | 444
  B Victoria | 36.3 [34.1 to 38.6] |  | 15.5 [12.3 to 19.3]
  B Yamagata: number analyzed (Participants) | 1751 | 437 | 0
  B Yamagata | 46.7 [44.3 to 49.0] | 17.4 [14.0 to 21.3] |
Statistical Analysis 1: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1); B Yamagata: The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction; Test type: Superiority — Superiority in seroconversion was observed if the lower limit of the 2-sided 95% CI of the difference of seroconversion rates between groups is > 10% for each applicable comparison; Difference in Percentage = 29.27, 95% CI 2-sided [24.78 to 33.29]
Statistical Analysis 2: Comparison: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) vs High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2); B Victoria: The 2-sided 95% CI for the difference was based on the Wilson score method without continuity correction; Test type: Superiority — [test comment as in outcome 5, analysis 1]; Difference in Percentage = 20.78, 95% CI 2-sided [16.5 to 24.61]

6. Secondary Outcome: Percentage of Participants Achieving Seroprotection Against Antigens Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: A/H1N1 (A1), A/H3N2 (A2), B Victoria lineage (B1), and B Yamagata lineage (B2). Seroprotection was defined as a HAI titer >=40 (1/dilution) at Day 0 and Day 28.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Analysis was performed on PPAS. Here, 'number analyzed' = participants with available data for each category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1680 | 423 | 430
percentage of participants
  A/H1N1: Day 0: number analyzed (Participants) | 1669 | 420 | 430
  A/H1N1: Day 0 | 69.4 [67.2 to 71.6] | 67.9 [63.2 to 72.3] | 70.1 [65.5 to 74.4]
  A/H3N2: Day 0: number analyzed (Participants) | 1668 | 420 | 430
  A/H3N2: Day 0 | 77.4 [75.3 to 79.4] | 78.1 [73.8 to 82.0] | 77.8 [73.6 to 81.7]
  B Victoria: Day 0: number analyzed (Participants) | 1669 | 421 | 430
  B Victoria: Day 0 | 88.9 [87.2 to 90.3] | 87.9 [84.4 to 90.8] | 88.8 [85.4 to 91.6]
  B Yamagata : Day 0: number analyzed (Participants) | 1669 | 421 | 430
  B Yamagata : Day 0 | 89.6 [88.0 to 91.0] | 88.1 [84.6 to 91.1] | 90.9 [87.8 to 93.4]
  A/H1N1: Day 28 | 95.1 [94.0 to 96.1] | 96.7 [94.5 to 98.2] | 95.6 [93.2 to 97.3]
  A/H3N2: Day 28: number analyzed (Participants) | 1679 | 423 | 430
  A/H3N2: Day 28 | 96.9 [96.0 to 97.7] | 96.9 [94.8 to 98.4] | 96.7 [94.6 to 98.2]
  B Victoria: Day 28 | 99.0 [98.5 to 99.5] | 99.1 [97.6 to 99.7] | 96.5 [94.3 to 98.0]
  B Yamagata : Day 28 | 99.3 [98.8 to 99.7] | 96.7 [94.5 to 98.2] | 99.1 [97.6 to 99.7]

7. Secondary Outcome: Geometric Mean Titers of Influenza Antibodies (Seroneutralization [SN] Assay) Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: GMTs of anti-influenza antibodies were measured using SN assay for 4 strains: A/H1N1 (A1), A/H3N2 (A2), B Victoria lineage (B1), and B Yamagata lineage (B2).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Expanded immunogenicity subset:participants who received at least 1 dose of trial vaccine& had post-vaccination blood sample HAI result for at least 1 strain& were randomized into expanded immunogenicity subset with at least 1 post-vaccination SN assay result for at least 1 strain.'Number analyzed'=participants with available data for each category
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 102 | 102 | 99
titers (1/dilution)
  A/H1N1: Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H1N1: Day 0 | 412 [306 to 555] | 427 [328 to 556] | 416 [311 to 555]
  A/H3N2: Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H3N2: Day 0 | 497 [417 to 592] | 536 [436 to 660] | 593 [493 to 715]
  B Victoria: Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Victoria: Day 0 | 458 [359 to 583] | 452 [367 to 556] | 430 [344 to 537]
  B Yamagata: Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Yamagata: Day 0 | 156 [124 to 196] | 155 [126 to 190] | 192 [152 to 242]
  A/H1N1: Day 28 | 2229 [1789 to 2776] | 2050 [1564 to 2687] | 1686 [1331 to 2135]
  A/H3N2: Day 28 | 1404 [1133 to 1741] | 1327 [1056 to 1667] | 1301 [1070 to 1583]
  B Victoria: Day 28 | 1288 [1055 to 1573] | 1114 [916 to 1354] | 590 [476 to 730]
  B Yamagata: Day 28 | 546 [438 to 682] | 259 [207 to 325] | 494 [390 to 626]

8. Secondary Outcome: GMTRs of Influenza Antibodies (SN Assay) Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: GMTRs of anti-influenza antibodies were measured using SN assay for 4 strains: A/H1N1 (A1), A/H3N2 (A2), B Victoria lineage (B1), and B Yamagata lineage (B2). GMTRs were calculated as the ratio of GMTs post vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Analysis was performed on expanded immunogenicity subset. Here, 'number analyzed' = participants with available data for each category.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 102 | 102 | 99
ratio
  A/H1N1: Day28/Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H1N1: Day28/Day 0 | 5.40 [3.90 to 7.48] | 5.05 [3.86 to 6.60] | 4.06 [3.17 to 5.18]
  A/H3N2: Day28/Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H3N2: Day28/Day 0 | 2.83 [2.31 to 3.46] | 2.50 [2.04 to 3.06] | 2.19 [1.80 to 2.67]
  B Victoria: Day28/Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Victoria: Day28/Day 0 | 2.81 [2.21 to 3.58] | 2.47 [2.04 to 2.99] | 1.37 [1.16 to 1.62]
  B Yamagata: Day28/Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Yamagata: Day28/Day 0 | 3.51 [2.80 to 4.39] | 1.66 [1.41 to 1.95] | 2.58 [2.18 to 3.05]

9. Secondary Outcome: Number of Participants With Neutralization Antibody Titers at Day 0 and Day 28
Description: Neutralizing Antibody titer was measured for each influenza strain with the SN method for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). Neutralizing antibody was defined as titers >=20 (1/dilution), >=40 (1/dilution), >=80 (1/dilution) at Day 0 and Day 28.
Time Frame: Day 0, Day 28
Population: Analysis was performed on expanded immunogenicity subset.
Measure: Count of Participants; unit: Participants
Groups:
- High-Dose Quadrivalent Influenza Vaccine (QIV-HD): Participants randomized to receive a single injection of the high dose QIV-HD by IM route at Day 0.
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 102 | 102 | 99
Participants
  A/H1N1: >=20 (1/dil): Day 0 | 97 | 99 | 98
  A/H1N1: >=40 (1/dil): Day 0 | 95 | 96 | 91
  A/H1N1: >=80 (1/dil): Day 0 | 89 | 89 | 84
  A/H3N2: >=20 (1/dil): Day 0 | 102 | 100 | 99
  A/H3N2: >=40 (1/dil): Day 0 | 102 | 100 | 99
  A/H3N2: >=80 (1/dil): Day 0 | 99 | 100 | 98
  B Victoria: >=20 (1/dil): Day 0 | 101 | 100 | 99
  B Victoria: >=40 (1/dil): Day 0 | 97 | 99 | 99
  B Victoria: >=80 (1/dil): Day 0 | 91 | 96 | 93
  B Yamagata: >=20 (1/dil): Day 0 | 98 | 98 | 99
  B Yamagata: >=40 (1/dil): Day 0 | 91 | 93 | 87
  B Yamagata: >=80 (1/dil): Day 0 | 75 | 75 | 74
  A/H1N1: >=20 (1/dil): Day 28 | 102 | 102 | 99
  A/H1N1: >=40 (1/dil): Day 28 | 102 | 102 | 99
  A/H1N1: >=80 (1/dil): Day 28 | 102 | 100 | 99
  A/H3N2: >=20 (1/dil): Day 28 | 102 | 102 | 99
  A/H3N2: >=40 (1/dil): Day 28 | 102 | 102 | 99
  A/H3N2: >=80 (1/dil): Day 28 | 102 | 101 | 99
  B Victoria: >=20 (1/dil): Day 28 | 102 | 102 | 99
  B Victoria: >=40 (1/dil): Day 28 | 102 | 102 | 99
  B Victoria: >=80 (1/dil): Day 28 | 102 | 102 | 97
  B Yamagata: >=20 (1/dil): Day 28 | 102 | 101 | 99
  B Yamagata: >=40 (1/dil): Day 28 | 102 | 99 | 97
  B Yamagata: >=80 (1/dil): Day 28 | 99 | 83 | 91

10. Secondary Outcome: Number of Participants With Two-Fold and Four-Fold Increase in Neutralization Antibody Titer at Day 28
Description: Neutralizing Antibody titer was measured for each influenza strain with the SN method for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). 2-fold and 4-fold rise was defined as the computed value = post-vaccination computed value / baseline computed value.
Time Frame: Day 28
Population: Analysis was performed on expanded immunogenicity subset. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 102 | 100 | 99
Participants
  Participants With 2-Fold Rise: A/H1N1 | 74 | 71 | 64
  Participants With 4-Fold Rise: A/H1N1 | 43 | 50 | 41
  Participants With 2-Fold Rise: A/H3N2 | 52 | 48 | 42
  Participants With 4-Fold Rise: A/H3N2 | 27 | 24 | 23
  Participants With 2-Fold Rise: B Victoria | 52 | 51 | 24
  Participants With 4-Fold Rise: B Victoria | 28 | 23 | 8
  Participants With 2-Fold Rise: B Yamagata | 65 | 31 | 55
  Participants With 4-Fold Rise: B Yamagata | 36 | 11 | 29

11. Secondary Outcome: Number of Participants With Detectable Neutralization Antibody Titers at Day 0 and Day 28
Description: Neutralizing Antibody titer was measured for each influenza strain with the SN method for 4 strains: A/H1N1, A/H3N2, B Victoria lineage (B1), and B Yamagata lineage (B2). Detectable neutralization antibody titer >= 1:10 (1/dilution) at Day 0 and Day 28.
Time Frame: Day 0, Day 28
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 102 | 102 | 99
Participants
  A/H1N1: Titer >= 1:10: Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H1N1: Titer >= 1:10: Day 0 | 100 | 100 | 99
  A/H1N1: Titer >= 1:10: Day 28 | 102 | 102 | 99
  A/H3N2: Titer >= 1:10: Day 0: number analyzed (Participants) | 102 | 100 | 99
  A/H3N2: Titer >= 1:10: Day 0 | 102 | 100 | 99
  A/H3N2: Titer >= 1:10: Day 28 | 102 | 102 | 99
  B Victoria: Titer >= 1:10: Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Victoria: Titer >= 1:10: Day 0 | 102 | 100 | 99
  B Victoria: Titer >= 1:10: Day 28 | 102 | 102 | 99
  B Yamagata: Titer >= 1:10: Day 0: number analyzed (Participants) | 102 | 100 | 99
  B Yamagata: Titer >= 1:10: Day 0 | 100 | 100 | 99
  B Yamagata: Titer >= 1:10: Day 28 | 102 | 102 | 99

12. Secondary Outcome: Number of Participants Reporting Solicited Injection-site and Systemic Reactions Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or High-Dose Trivalent Influenza Vaccine
Description: Solicited injection site: Pain, Erythema, Swelling, Induration, and Bruising. Grade 3 reactions: Pain - interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention; Erythema, Swelling, Induration, and Bruising: >100 millimeters (mm). Systemic reactions: Fever, Headache, Malaise, Myalgia, and Shivering. Grade 3 reactions: Fever: >=39°C; Headache, Malaise, Myalgia, and Shivering: interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on safety analysis set that included all participants who had received study vaccine. All participants had their safety analyzed according to the vaccine they actually received. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1777 | 443 | 450
Participants
  Fever: Any Grade: number analyzed (Participants) | 1761 | 437 | 448
  Fever: Any Grade | 7 | 3 | 5
  Fever: Grade 3: number analyzed (Participants) | 1761 | 437 | 448
  Fever: Grade 3 | 3 | 1 | 1
  Headache: Any Grade: number analyzed (Participants) | 1768 | 440 | 449
  Headache: Any Grade | 254 | 63 | 58
  Headache: Grade 3: number analyzed (Participants) | 1768 | 440 | 449
  Headache: Grade 3 | 11 | 2 | 2
  Malaise: Any Grade: number analyzed (Participants) | 1768 | 440 | 449
  Malaise: Any Grade | 233 | 52 | 67
  Malaise: Grade 3: number analyzed (Participants) | 1768 | 440 | 449
  Malaise: Grade 3 | 13 | 3 | 1
  Myalgia: Any Grade: number analyzed (Participants) | 1768 | 440 | 449
  Myalgia: Any Grade | 402 | 80 | 88
  Myalgia: Grade 3: number analyzed (Participants) | 1768 | 440 | 449
  Myalgia: Grade 3 | 16 | 3 | 3
  Shivering: Any Grade: number analyzed (Participants) | 1768 | 440 | 449
  Shivering: Any Grade | 95 | 20 | 22
  Shivering: Grade 3: number analyzed (Participants) | 1768 | 443 | 449
  Shivering: Grade 3 | 5 | 3 | 0
  Injection Site Bruising: Any: number analyzed (Participants) | 1765 | 439 | 448
  Injection Site Bruising: Any | 23 | 6 | 4
  Injection Site Bruising: Grade 3: number analyzed (Participants) | 1765 | 439 | 448
  Injection Site Bruising: Grade 3 | 0 | 0 | 0
  Injection Site Erythema: Any: number analyzed (Participants) | 1768 | 440 | 449
  Injection Site Erythema: Any | 110 | 30 | 21
  Injection Site Erythema: Grade 3: number analyzed (Participants) | 1768 | 440 | 449
  Injection Site Erythema: Grade 3 | 11 | 1 | 1
  Injection Site Induration: Any: number analyzed (Participants) | 1766 | 439 | 448
  Injection Site Induration: Any | 66 | 17 | 14
  Injection Site Induration: Grade 3: number analyzed (Participants) | 1766 | 439 | 448
  Injection Site Induration: Grade 3 | 3 | 0 | 1
  Injection Site Pain: Any: number analyzed (Participants) | 1768 | 440 | 449
  Injection Site Pain: Any | 731 | 172 | 152
  Injection Site Pain: Grade 3: number analyzed (Participants) | 1768 | 440 | 449
  Injection Site Pain: Grade 3 | 12 | 1 | 1
  Injection Site Swelling: Any: number analyzed (Participants) | 1766 | 439 | 448
  Injection Site Swelling: Any | 86 | 23 | 19
  Injection Site Swelling: Grade 3: number analyzed (Participants) | 1766 | 439 | 448
  Injection Site Swelling: Grade 3 | 5 | 0 | 1

13. Secondary Outcome: Number of Participants With Immediate Adverse Event (AEs)
Description: Participants were observed for 30 minutes after vaccination, and any unsolicited systemic AEs occurring during that time was recorded as immediate unsolicited systemic AEs (AEs that were related to the investigational product) in the case report book (CRB). Unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of symptom and/ or onset post-vaccination. Unsolicited AEs included both serious and non-serious unsolicited AEs. A serious adverse event was any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: Within 30 minutes after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1777 | 443 | 450
Participants | 5 | 0 | 2

14. Secondary Outcome: Number of Participant With Unsolicited Adverse Event (AE)
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of symptom and/or onset post-vaccination. Unsolicited AEs included both serious and non-serious unsolicited AEs. A serious adverse event was any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event.
Time Frame: Within 28 days after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1777 | 443 | 450
Participants | 292 | 79 | 68

15. Secondary Outcome: Number of Participant With Serious Adverse Event
Description: An serious adverse event was any untoward medical occurrence that at any dose results in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity,is a congenital anomaly/birth defect, or was an important medical event.
Time Frame: Up to 6 months after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
Number analyzed (Participants) | 1777 | 443 | 450
Participants | 80 | 29 | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 (post-vaccination) up to 28 days after last vaccination. Solicited Reaction (SR) data were collected up to Day 7 after each vaccination. Serious adverse event data were collected throughout the study (up to 180 days after last vaccination).
Description: Analysis was performed on safety analysis set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Groups:
- High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1): Participants randomized to receive a single injection of the licensed high dose TIV-HD1 by IM route at Day 0.
- High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2): Participants randomized to receive a single injection of the investigational TIV-HD2 by IM route at Day 0.
Arm/Group | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2)
All-Cause Mortality (participants affected / at risk) | 3/1777 | 2/443 | 0/450
Serious Adverse Events (participants affected / at risk) | 80/1777 | 29/443 | 19/450
Other Adverse Events (participants affected / at risk) | 935/1777 | 234/443 | 206/450
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) (N=1777) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) (N=443) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2) (N=450)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 1 (1) | 1 (2)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular Stent Thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae Viral Laryngotracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 2 (3) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Small Fibre Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Stenosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Quadrivalent Influenza Vaccine (QIV-HD) (N=1777) | High-Dose Trivalent Influenza Vaccines (Licensed TIV-HD1) (N=443) | High-Dose Trivalent Influenza Vaccine(Investigational TIV-HD2) (N=450)
Chills (General disorders) | 96 (97) | 20 (20) | 22 (22)
Injection Site Erythema (General disorders) | 110 (112) | 30 (31) | 21 (21)
Injection Site Pain (General disorders) | 731 (731) | 172 (172) | 152 (152)
Injection Site Swelling (General disorders) | 86 (87) | 23 (23) | 19 (19)
Malaise (General disorders) | 233 (234) | 52 (53) | 67 (67)
Myalgia (Musculoskeletal and connective tissue disorders) | 404 (404) | 81 (81) | 88 (88)
Headache (Nervous system disorders) | 258 (262) | 65 (65) | 59 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable partcipant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03282240/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03282240/SAP_001.pdf